CLINICAL TRIAL: NCT03865901
Title: Subject Enrollment and Specimen Collection Protocol to Validate the Performance of the Mellitus GCD59 ELISA for Gestational Diabetes Screening
Brief Title: Protocol to Validate the Performance of the Mellitus Glycated CD59 ELISA for Gestational Diabetes Screening
Status: Withdrawn | Type: Observational
Why Stopped: Further product development is needed prior to clinical study testing
Sponsor: Mellitus, LLC (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Other Study IDs: CSP-MEL-002
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Gestational Diabetes
Keywords: in vitro diagnostic; GDM; gestational diabetes mellitus; screening; pregnancy; prenatal care; women's health
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Non-diabetic pregnant women: Non-diabetic women with singleton pregnancy undergoing screening for gestational diabetes who provide plasma samples for testing with the Mellitus GCD59 Test
  Interventions: Diagnostic Test: Mellitus GCD59 Test

INTERVENTIONS:
Diagnostic Test: Mellitus GCD59 Test — An ELISA for screening for the risk of gestational diabetes
  Other Names: Mellitus GCD59 ELISA

SUMMARY:
Demonstrate effective performance of the Mellitus GCD59 Test (an ELISA) in screening for gestational diabetes mellitus (GDM)

DETAILED DESCRIPTION:
Validate the performance of the Mellitus GCD59 ELISA as a screening test for GDM by evaluating its negative predictive value (NPV) and positive predictive value (PPV) to identify pregnant women at risk for GDM. Sensitivity and specificity of the Mellitus GCD59 ELISA will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older at enrollment
2. Has an established viable singleton pregnancy
3. Is recommended for routine GDM screening between 24-28 weeks gestation
4. Has confirmed gestational age of 24-28 weeks at the Screening Visit
5. Is willing and able to provide documentation of informed consent

Exclusion Criteria:

1. Has diabetes before pregnancy or has already been diagnosed with GDM
2. Has contraindications for drinking oral glucose solution up to 100 g of sugar
3. Is taking metformin for any reason
4. Has any concomitant illness, disease or condition that, in the clinical judgment of the investigator, is likely to prevent the subject from complying with any aspect of the protocol, or that may put the subject at unacceptable risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — non-diabetic pregnant women
Study Population: Nondiabetic women with a singleton pregnancy recommended for routine GDM screening between 24-28 weeks gestation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) and positive predictive value (PPV) of the Mellitus GCD59 ELISA for gestational diabetes mellitus screening | The 24-28th gestational week of singleton pregnancy
  NPV and PPV will be based on two or more abnormal oral glucose tolerance test (OGTT) results (abnormal for OGTT as defined by Carpenter and Coustan diagnostic criteria)

SECONDARY OUTCOMES:
Sensitivity and specificity of the Mellitus GCD59 ELISA for gestational diabetes mellitus screening, using two or more abnormal OGTT results (abnormal for OGTT as defined by Carpenter and Coustan diagnostic criteria) | The 24-28th gestational week of singleton pregnancy
NPV, PPV, sensitivity and specificity of the GCD59 ELISA for the risk of GDM using one or more abnormal OGTT results | The 24-28th gestational week of singleton pregnancy
Sensitivity and specificity of the GCD59 ELISA to that of glucose load test (GLT) using two or more abnormal oral glucose tolerance test (OGTT) results | The 24-28th gestational week of singleton pregnancy

OTHER OUTCOMES:
Negative predictive value (NPV) and positive predictive value (PPV) of the GCD59 ELISA for a range of gestational diabetes mellitus (GDM) prevalence values likely to be encountered in clinical practice in the United States | The 24-28th gestational week of singleton pregnancy
Sensitivity and specificity of the GCD59 ELISA across relevant subgroups | The 24-28th gestational week of singleton pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A Lonergan, Study Chair — Mellitus, LLC
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - UC Irvine Health, Orange, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Christina Care Health System, Newark, Delaware
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - UMass Medical School/UMass Memorial Health Care, Worcester, Massachusetts
  - Spectrum Hleath, Grand Rapids, Michigan
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University School of Medicine, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Austin Maternal-Fetal Medicine, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No